CLINICAL TRIAL: NCT06720428
Title: Development of a Prototype of Acupoint Therapy Device for Dry Eye and Preliminary Verification of Its Clinical Efficacy
Brief Title: Acupoint Therapy Device for Dry Eye
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Jing Yu, Director, Ophthalmology, Clinical Professor, Shanghai 10th People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YNCR2B003
Record Dates: First submitted 2024-08-28; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Dry Eye
Keywords: Acupuncture treatment; Dry Eye Acupoint Therapeutic Instrument; Safety; Validity
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Lubricant Eye Drops

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dry eye acupoint therapy instrument treatment group One (Experimental): Dry eye acupoint therapy instrument treatment group One was treated with instrument twice a week, at least two day apart, each time lasting 30 minutes. Treatment points include Jingming, Cunzhu, Si Zhukong , Sun , Sibai and Chengqi.
  Interventions: Device: dry eye acupoint therapy instrument; Drug: Artificial tear
- Dry eye acupoint therapy instrument treatment group Two (Experimental): Dry eye acupoint therapy instrument treatment group Two had the same treatment method with different treatment parameters.
  Interventions: Device: dry eye acupoint therapy instrument; Drug: Artificial tear
- Artificial tear treatment group (Active Comparator): The artificial tear treatment group was treated with artificial tear (Ali eye drops) four times a day.
  Interventions: Drug: Artificial tear

INTERVENTIONS:
Device: dry eye acupoint therapy instrument — The dry eye acupuncture point treatment device treat dry eye through stimulating acupuncture points by low pulse current.
  Arms: Dry eye acupoint therapy instrument treatment group One; Dry eye acupoint therapy instrument treatment group Two
Drug: Artificial tear — 0.3% Ali eye drops

SUMMARY:
To built a dry eye acupoint therapeutic instrument by stimulating acupoints with low impulse current .And the safety of the dry eye acupoint treatment device will be tested and the initial validation will be verified.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who meet the diagnostic criteria for dry eye: The diagnostic and classification criteria refer to the Consensus of Chinese dry eye Experts: Definition and Classification (2020);
2. this study included patients with dry eyes can be treated as usual or are using artificial tears, also can be never accepted artificial tears treatment;
3. this research project, informed consent and signed informed consent form, participants are willing to accept treatment.

Those who met the above criteria could be included in the study.

Exclusion Criteria:

1. Patients with other eye diseases, acute inflammation or allergy of the eye or skin around the eye: such as blepharitis, lacrimal duct obstruction, congenital absence or dysplasia of lacrimal gland, anterior ganglia inflammation, such as trachoma, chemical burn and other corneal and conjunctival lesions, extensive scar of the eyelid conjunctival, long-term use of anti-glaucoma eye drops for glaucoma;
2. Those who have undergone external or internal eye surgery in the past 6 months；
3. Patients who have undergone tear punctum embolization or submandibular gland transplantation;
4. Wearing contact lenses within the past 3 months； （5）History of ocular trauma; （6）Active fundus lesions in the past 3 months； （7）People who are allergic to artificial tears; （8）Suffering from diseases that affect tear secretion, such as facial paralysis, diabetes, and hyperthyroidism;

(9)Patients with serious life-threatening primary diseases such as cardiovascular, cerebrovascular, liver, kidney, and hematopoietic system diseases, as well as mental illness; (10)Attending other clinical trials.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Schirmer's test (SLT) | baseline and 8 weeks post-treatment
  The Schirmer test uses filter paper to wick up tears and measure the amount of production.
Tear film breakup time (TBUT) | baseline and 8 weeks post-treatment
  The time interval between keeping eyes open after blinking until the first dry spot appears on the tear film surface is one of the important criteria to evaluate the stability of tear film.
Ocular Surface Disease Index, OSDI | baseline and 8 weeks post-treatment
  The most commonly used questionnaire in clinical diagnosis of dry eye. It is mainly used to diagnose dry eye and assess the severity of the condition
Corneal fluorescein staining (CFS) | baseline and 8 weeks post-treatment
  Corneal fluorescein staining (CFS) is a valuable clinical tool to assess the viability of the epithelium.

SECONDARY OUTCOMES:
MGD | baseline and 8 weeks post-treatment
  Meibomian Gland (MG) expressibility and secretion quality

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality, China